CLINICAL TRIAL: NCT03211663
Title: A Prospective, Multi-Center Study To Assess Performance of MOTO Medial® in Unicompartmental Knee Arthroplasty (UKA).
Brief Title: Performance of MOTO Medial® Unicompartmental Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MUSA-K-MTM-001
Record Dates: First submitted 2017-06-28; First posted 2017-07-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interventional : MOTO Medial® UKA: Interventional : Patients who are planned to undergo a primary medial UKA using the MOTO Medial® will be enrolled.
  Interventions: Device: MOTO Medial® UKA

INTERVENTIONS:
Device: MOTO Medial® UKA — Knee replacement surgery with the MOTO Medial® UKA
  Other Names: Medial Unicondylar Knee Replacement

SUMMARY:
This is a prospective, multi-center study, designed to assess mid-term performance of the MOTO Medial® Unicompartmental Knee Arthroplasty (UKA), with patient report outcomes, clinical findings and radiographic analysis.

DETAILED DESCRIPTION:
This is a prospective, multi-center study, designed to assess mid-term performance of the MOTO Medial® UKA, with patient report outcomes, clinical findings and radiographic analysis. Additionally, several perioperative factors, medical and surgical history will be evaluated. Implant survival and complications will be detailed throughout the study. Data from pre-operative evaluation, day of surgery, and post-operatively at 4 weeks, 6 months, and years 1, 2 & 5, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF).

  * Ability to understand and provide written authorization for use and disclosure of personal health information.
  * Subject who are able and willing to comply with the study protocol and follow-up visits.
  * Must be 18 years or older to participate.
  * Subjects must have medial knee disease in the affected knee compliant with the FDA-approved indications for use of MOTO Medial® UKA.
  * Must have had no prior arthroplasty to the medial compartment of the study knee.
  * Subjects must be able to return for the follow-up appointments, and have the mental capacity to cooperate and complete Patient Reported Outcome questionnaires, physical exam and radiographs.

Exclusion Criteria:

* Knee ligament instability (deficiency of cruciate or collateral ligaments)

  * Inflammatory Arthritis
  * History of prior knee infection
  * History of Alcoholism or Drug Abuse
  * Currently on chemotherapy or radiation therapy for neoplastic disease. Medacta MOTO Medial® Version 1 Confidential Page 9 of 36 June 5, 2017
  * Currently on immunosuppressive medications including steroids
  * History of known sensitivity or allergy to materials used in orthopedic implants, specifically Titanium and Cobalt-Chrome alloys
  * Habitual use of narcotic pain medications prior to surgery (more than 3 doses or pills per week)
  * History of metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis (e.g., Osteomalacia, Ricketts)
  * History of chronic pain issues for reasons other than knee pain.
  * Women who are pregnant.
  * Psychiatric illness
  * Any patient, in the opinion of the investigator, is unable to fully comply with the surgical, rehabilitation, or follow-up aspects of this procedure.
  * Prior joint arthroplasty on the target knee, including prior medial UKA (revision), lateral UKA, or Patellofemoral Joint
  * Prior high tibial osteotomy (HTO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Knee Society Score Objective | Baseline, post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of improvement of clinical outcomes following knee replacement surgery using the Knee Society Score Questionnaire
Change from baseline in Knee Osteoarthritis Outcome Score | Baseline, post-operative 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of improvement of activity levels following knee replacement surgery using the Knee Osteoarthritis Score Questionnaire
Change from baseline in Forgotten Joint Score | post-operative 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of the improvement of joint specific outcomes following knee replacement surgery using the Forgotten Joint Score Questionnaire.
Knee Society Score | Baseline
  Assessment of pre-op expectations questionnaire
Change from baseline in Knee Society Score | post-operative 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of the improvement post-op satisfaction following knee replacement surgery using the Knee Society Score questionnaire.
Change from baseline in Veterans Rand 12 Score | Baseline, post-operative 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of the improvement of your health using the Veterans Rand 12 score questionnaire.
Change from baseline in Oxford Knee Score | Baseline, post-operative 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assessment of the improvement of knee function following knee replacement surgery using the Oxford Knee Score questionnaire.
Change from baseline in Medication for Osteoarthritis | Baseline, post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Documentation of osteoarthritis medications
Change from baseline in Knee Wound Assessment | post-operative 2-6 weeks, 4-8 months
  Assessment of wound drainage, swelling and infection in surgical knee
Change from baseline in Visual Analog Scale score | baseline, post-operative 2-6 weeks, 4-8 months
  Assessment of the improvement of patient knee pain following knee replacement surgery using the VAS score questionnaire.
Severity of osteoarthritis in the knee compartments | Baseline
  Determine by radiographic analysis for disease progression
Change from baseline in Knee Alignment | Baseline, post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Determine by radiographic analysis Varus or Valgus
Change from baseline of Implant position fixation | post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Determine by radiographic analysis by measuring Radio Lucent lines in millimeters.
Change from baseline of implant survivorship | post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Determine by radiographic analysis of bone fracture, implant fracture, fixation and wear

SECONDARY OUTCOMES:
Number of knee Implant faliures | post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Reoperations, revisions, removals, and device related adverse events
K & L Grading | Baseline
  Assessment of Osteoarthritis Disease Grade of the knee compartment
Age of patient | Baseline
  Date of birth (age)
Demographics | Baseline
  Height in inches, weight in pounds to determine BMI
Number of male or female patients | Baseline
  Gender description male or female
Occurrence of Knee Treatments prior to surgery | Baseline
  Prior treatments of knee such as bracing, medication, injections, arthroscopy, ligament and cartilage procedures
Occurrence of prior medical and surgical history | Baseline
  Medical and surgical history of patient prior to knee surgery
Post-operative pain medications | post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Medications after knee surgery
Return to Work/Activity questionnaire | post-operative 4-8 months, 9-15 months, 18-30 months
  Assessment of ability to return to work or other activities following surgery
Implant demographics | day of surgery
  Implant femoral and tibial size and poly thickness
Anesthetic | day of surgery
  type of anesthesia used during surgery
Estimated blood loss | day of surgery
  Volume of blood loss during surgery
Length of surgery | day of surgery
  Time in minutes of skin to skin
Length of Hospital Stay | day of surgery
  Length of stay in hours
Frequency of Facility type used for knee surgery | day of surgery
  Type of facility used for knee surgery
Tourniquet Time | day of surgery
  Tourniquet time in minutes
Complications | day of surgery, post-operative 2-6 weeks, 4-8 months, 9-15 months, 18-30 months and 51-69 months
  Assess adverse events and Serious adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Unova Health Clinic, Lady Lake, Florida
  - Ellis & Badenhausen Orthopaedics PSC, Louisville, Kentucky
  - Ortho Montana, Billings, Montana
  - Duke University, Durham, North Carolina
  - Whole Health Joint Replacement, Meadville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No